CLINICAL TRIAL: NCT00323362
Title: Phase II Study of Imatinib Mesylate and Gemcitabine for Recurrent/Metastatic Non-small Cell Lung Cancer (NSCLC)
Brief Title: Gemcitabine and Imatinib Mesylate in Treating Patients With Recurrent or Metastatic Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Toxicity
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000539557; P30CA072720 (NIH); 030503 (Other: CINJ); 0220060014 (Other: UMDNJ IRB); NJ1505 (Other: CINJ)
Record Dates: First submitted 2006-03-07; First posted 2006-05-09 (Estimated); Results first posted 2014-05-22 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-04

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine hydrochloride and imatinib mesylate (Experimental)
  Interventions: Drug: gemcitabine hydrochloride; Drug: imatinib mesylate

INTERVENTIONS:
Drug: gemcitabine hydrochloride — 1000 mg/m2 given intravenously at a FDR of 10 mg/m2/min on Days 3 and 10, every 21 days.
Drug: imatinib mesylate — 400 mg/day orally, given Days 1-5 and 8-12 every 21 days

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving gemcitabine together with imatinib mesylate may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with imatinib mesylate works in treating patients with recurrent or metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the response rate in patients with recurrent or metastatic non-small cell lung cancer treated with gemcitabine hydrochloride and imatinib mesylate.

Secondary

* Assess time to progression in patients treated with this regimen.
* Assess overall survival and 1-year survival of patients treated with this regimen.
* Assess the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter, nonrandomized, uncontrolled, open-label study.

Patients receive gemcitabine hydrochloride IV on days 3 and 10 and oral imatinib mesylate once daily on days 1-5 and 8-12. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 53 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell cancer

  * Recurrent disease after adjuvant treatment OR progressive disease after 1 prior treatment for recurrent or metastatic disease
* Received at least 1 prior chemotherapy regimen and meets the following criteria:

  * No more than 1 prior chemotherapeutic regimen in the recurrent or metastatic setting
  * Patients who received prior chemotherapy in the adjuvant setting are eligible when 1 of the following criteria is met:

    * In first recurrence (after 1 prior regimen)
    * Received first-line chemotherapy in the recurrent setting after 2 prior regimens
* Measurable disease

  * Must have ≥ 1 measurable target lesion outside prior radiotherapy field OR radiologic confirmation of disease progression within a prior radiotherapy field
* No known or untreated brain metastases or carcinomatous meningitis

  * Clinically stable, treated brain metastases allowed provided it has been > 7 days since prior steroids

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 3 months
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* Able to swallow oral medication
* No concurrent medical condition that would preclude study compliance
* No history of allergic reaction to compounds of similar chemical or biological composition to gemcitabine hydrochloride or imatinib mesylate
* No uncontrolled illness that would preclude study compliance, including any of the following:

  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia requiring therapy
  * Myocardial infarction within the past 6 months
  * Active infection
* No New York Heart Association class III-IV congestive heart failure
* No chronic liver disease (i.e., chronic active hepatitis, cirrhosis)
* No HIV positivity
* No other primary malignancies within the past 5 years, except carcinoma in situ of the cervix or nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* At least 3 weeks since prior anti-vascular endothelial growth factor therapy and recovered
* At least 3 weeks since prior radiotherapy and recovered
* More than 28 days since prior and no other concurrent investigational or commercial agents
* More than 2 weeks since prior major surgery
* No prior gemcitabine hydrochloride or imatinib mesylate for metastatic disease
* No prior tyrosine kinase inhibitor, except for gefitinib or erlotinib hydrochloride
* No concurrent therapeutic warfarin (prophylactic warfarin therapy ≤ 1 mg daily allowed)
* No other concurrent medications that would preclude study compliance
* No concurrent chronic systemic corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mika Sovak, MD, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (3):
- United States (3):
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seventeen patients were enrolled from April 2006 through October 2007 at Rutgers Cancer Institute of New Jersey, a comprehensive cancer cancert, and two of its affiliate hospitals within the CINJ Oncology Group.
Groups:
- Gemcitabine Hydrochloride and Imatinib Mesylate: gemcitabine hydrochloride : 1000 mg/m2 given intravenously at a FDR of 10 mg/m2/min on Days 3 and 10, every 21 days.
  imatinib mesylate : 400 mg/day orally, given Days 1-5 and 8-12 every 21 days
Period: Overall Study
Arm/Group | Gemcitabine Hydrochloride and Imatinib Mesylate
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine Hydrochloride and Imatinib Mesylate
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Meet Critieria for Response
Description: Response is considered Partial Response or Complete Response as per RECIST criteria.
  Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
  Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: 2 years
Population: Fourteen subjects were evaluable for response. Three subjects were not assessed.
Measure: Number; unit: percentage of patients who responded
Arm/Group | Gemcitabine Hydrochloride and Imatinib Mesylate
Number analyzed (Participants) | 14
percentage of patients who responded | 0

2. Secondary Outcome: Time to Progression
Time Frame: 2 years
Population: The study was closed early due to toxicity and insufficient data were collected to analyze this outcome measure.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Gemcitabine Hydrochloride and Imatinib Mesylate
Number analyzed (Participants) | 14
months | 2.77 (2.07)

3. Secondary Outcome: 1-year Survival
Description: Accrual duration is 2 years with an additional year for assessment of 1-year survival. Outcome measure time frame is about 3 years.
Time Frame: 3 years
Population: The study was closed early due to toxicity and insufficient data were collected to analyze this outcome measure.
Measure: Number; unit: percentage of patients
Arm/Group | Gemcitabine Hydrochloride and Imatinib Mesylate
Number analyzed (Participants) | 17
percentage of patients | 35

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Gemcitabine Hydrochloride and Imatinib Mesylate
Serious Adverse Events (participants affected / at risk) | 10/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine Hydrochloride and Imatinib Mesylate (N=17)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory - Nose (Vascular disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Death not associated with CTCAE term - Disease progression NOS (General disorders) | 4 (4)
Other toxicity (General disorders) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Skin (cellulitis) (Infections and infestations) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine Hydrochloride and Imatinib Mesylate (N=17)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 11 (27)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 11 (30)
Platelets (Blood and lymphatic system disorders) | 9 (13)
Hemoglobin (Blood and lymphatic system disorders) | 8 (15)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 9 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 8 (9)
Insomnia (General disorders) | 2 (2)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1)
Weight loss (General disorders) | 1 (1)
Pain - Bone (General disorders) | 4 (4)
Pain - Head/headache (General disorders) | 2 (3)
Pain - Muscle (General disorders) | 2 (3)
Pain - Back (General disorders) | 1 (1)
Pain - Extremity-limb (General disorders) | 1 (1)
Pain - Joint (General disorders) | 1 (1)
Pain - other (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (7)
Constipation (Gastrointestinal disorders) | 2 (3)
Anorexia (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Skin (cellulitis) (Infections and infestations) | 2 (2)
Infection - Other (Infections and infestations) | 1 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 1 (1)
Infection with unknown ANC - Skin (cellulitis) (Infections and infestations) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Mood alteration - Anxiety (Psychiatric disorders) | 1 (1)
Mood alteration - Depression (Psychiatric disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory - Nose (Vascular disorders) | 2 (2)
Hemorrhage, pulmonary/upper respiratory - Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemorrhage/Bleeding - Other (Vascular disorders) | 1 (2)
Edema: limb (Blood and lymphatic system disorders) | 3 (7)
Bladder spasms (Renal and urinary disorders) | 1 (1)
Incontinence, urinary (Renal and urinary disorders) | 1 (1)
Renal/Genitourinary - Other (Renal and urinary disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Death not associated with CTCAE term - Disease progression NOS (General disorders) | 1 (1)
Potassium, serum-low (hypokalemia) (Investigations) | 1 (1)
Vascular - Other (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The CINJ PI, and all co-authors, prior to submission or use, must review any abstract or manuscript.